CLINICAL TRIAL: NCT07395986
Title: A Multicenter, Randomized, Double-Masked, Placebo-Controlled Pilot Study to Evaluate the Efficacy and Safety of ZOC2017217 in Subjects With Age-Related Cataract
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Ocusun Ophthalmic Pharmaceutical (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GOCS-H101-E06
Record Dates: First submitted 2026-01-15; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Age Related Cataracts
Keywords: Cataract; Cataracts; Age related cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control (Placebo Comparator): Drug with no active ingredients
  Interventions: Drug: Control
- Active (Experimental): ZOC2017217
  Interventions: Drug: 0.4% ZOC2017217

INTERVENTIONS:
Drug: 0.4% ZOC2017217 — Active Investigational Product
  Arms: Active
Drug: Control — Control
  Arms: Control

SUMMARY:
This is a multicenter, randomized, double-masked, placebo-controlled pilot study conducted in the United States (US) in subjects with age-related cataract in one or both eyes.

Approximately 40 subjects with age-related cataract will be stratified by race and Best Corrected Distance Visual Acuity (BCDVA) and randomized (1:1) to active investigational product (IP) or placebo.

Subjects will administer their assigned IP in the qualifying eye(s) two times a day (BID) for 24 weeks before being exited from the study. Subjects with new or ongoing ocular adverse events (AEs) at the time of planned study exit will be asked to return 2 weeks later for a safety follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  1. Are ≥50 years of age.
  2. Willing and able to provide informed consent and provide relevant privacy authorization(s).
  3. Willing and able to comply with study requirements and visit schedule.
  4. Able to successfully administer ophthalmic solution or have an appropriate designee (e.g., family member, health care professional) who can administer ophthalmic solution.

  6. Have calculated baseline BCDVA at Visit 2 (Randomization; Baseline; Day 1) that simultaneously meets Randomization Criteria.

  7. Have, in the opinion of the Investigator, age-related cataract (cortical, nuclear, posterior, mixed) in one or both eyes, as assessed using digital imaging after adequate mydriasis.

A. C < 5.0 B. N < 5.0 (both nuclear opalescence [NO] and nuclear color [NC]) C. P < 1.0 8. Have, in the opinion of the Investigator, sufficiently clear ocular media and adequate pupillary dilation to permit quality fundus imaging.

Exclusion Criteria:

* Ocular Exclusion Criteria:

Study Eye:

1. Have a history of ocular trauma.
2. Have a history of intraocular surgery, laser treatment, or corneal surgery. Note: Corneal refractive surgery more than 2 years prior to Visit 1 (Screening) is allowed.
3. Have, in the opinion of the Investigator, a cataract other than age-related cataract (e.g., traumatic, concurrent, metabolic, drug and toxic, radiation).
4. Have, in the opinion of the Investigator, any ocular disease or condition that is not stably controlled or is likely to affect central vision, including but not limited to:

   Glaucoma Elevated IOP (e.g., ≥30 mmHg) Optic neuropathy Age-related macular degeneration Diabetic retinopathy Retinal artery or vein occlusion Macular hole Retinal detachment Epiretinal membrane involving the fovea High myopia (i.e., spherical equivalent of subjective refraction ≥ -7.0 D) High hyperopia (i.e., spherical equivalent of subjective refraction > +4.00 D)
5. Have overall CFS >3.
6. Have active eye infection or inflammation, including but not limited to conjunctivitis, keratitis, scleritis, or endophthalmitis.

   Note: Mild inflammation (CFS <3 on the NEI scale) from ocular surface disease, including dry eye disease, is allowed.

   Non-study Eye:
7. Have high-contrast BCDVA under photopic conditions ≤19 letters.

   Either Eye:
8. Have a history of cataract surgery or be planning to undergo cataract surgery during the study.
9. Have newly developed or not stably controlled uveitis within the 6 months prior to Visit 1 (Screening).
10. Unwilling or unable to discontinue wearing contact lenses 14 days prior to Visit 2 (Randomization; Baseline; Day 1), and during the study conduct.
11. Requires, is likely to require, or is unwilling to discontinue the use of prohibited medications or procedures within 14 days prior to Visit 1 (Screening), or during the study conduct.

    A. Other ocular surgeries that may affect visual function, including but not limited to photodynamic therapy. B. Desferrioxamine, hydroxychloroquine, chloroquine, tamoxifen, phenothiazines, ethambutol, or other agents known to cause crystalline lens, retinal, or optic nerve toxicity.

    C. Chlorpromazine or corticosteroids that may aggravate crystalline lens opacity.

    Note: Topical non-ocular corticosteroids are allowed.

    General Exclusion Criteria:
12. Have a severe or not stably controlled systemic disease that may interfere with study participation or confound interpretability (e.g., acute phase of chronic obstructive pulmonary disease; congestive heart failure; severe hepatic or renal insufficiency; malignant tumors currently being treated with chemotherapy).
13. Have diabetes mellitus with HbA1c ≥7.5%.
14. Have hypertension that is not stably controlled at Visit 1 (Screening) A. Systolic blood pressure: >180 mmHg B. Diastolic blood pressure: >100 mmHg after standard of care
15. Have participated or are planning to participate in a clinical study for an investigational drug/medical device within 30 days prior to Visit 1 (Screening), or during the study conduct.
16. Are pregnant, nursing, or planning a pregnancy during the study.
17. Unwilling or unable to use an acceptable method of contraception throughout the study if a woman of childbearing potential (WOCBP).
18. Unwilling or unable to use an acceptable method of contraception throughout the study if a male sexual partner of a WOCBP.
19. Have a family member or household member enrolled in the study.
20. Have any condition, in the opinion of the Investigator, that makes the subject unsuitable for study participation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
BCDVA | Baseline as compared to Weeks 4, 12, and 24.
  Change from baseline in BCDVA at Weeks 4, 12, and 24.
Contrast Sensitivity | Baseline as compared to Weeks 4, 12, and 24.
  Change from baseline in contrast sensitivity at Weeks 4, 12, and 24.
Visual Function Questionnaire (VFQ-25) | Baseline compared to Weeks 4, 12, and 24.
  Change from baseline in Visual Function Questionnaire (VFQ-25) scores at Weeks 4, 12, and 24. VFQ-25 score total should increase from the baseline visit to show better visual function at Weeks 4, 12, and 24.
Crystalline Lens Opacity | Baseline compared to Weeks 4, 12, and 24.
  Change from baseline in crystalline lens opacity at Weeks 4, 12, and 24.
BCDVA | Baseline compared to Weeks 4, 12, and 24.
  Proportion of subjects gaining ≥5, ≥10, or ≥15 letters from baseline in BCDVA at Weeks 4, 12, and 24.
BCDVA | Baseline compared to Weeks 4, 12, and 24.
  Proportion of subjects losing ≤5, ≤10, or ≤15 letters from baseline in BCDVA at Weeks 4, 12, and 24.
BCDVA | Baseline compared to Weeks 4, 12, and 24.
  Proportion of subjects achieving BCDVA ≥0.3, 0.1, or 0.0 Logarithm of the Minimum Angle of Resolution (LogMAR; Snellen: 20/40, 20/25, or 20/20) at Weeks 4, 12, and 24.

SECONDARY OUTCOMES:
Safety, AEs | From the start of use of the IP at Visit 2 (Day 1) to the time the subject is exited after Visit 6 procedures and assessments are conducted. Visit 6 is conducted 2 weeks after the last dose is given at Week 24.
  AE monitoring (ocular and non-ocular)
Safety, Clinically Relevant Changes | From the start of use of the IP at Visit 2 (Day 1) to the time the subject is exited after Visit 6 procedures and assessments are conducted. Visit 6 is conducted 2 weeks after the last dose is given at Week 24.
  Clinically relevant changes from baseline in the following:
  Vital signs Slit-lamp biomicroscopy Corneal fluorescein staining (CFS)-National Eye Institute (NEI) Grading Scale Corneal endothelial cell count Intraocular pressure (IOP) Dilated fundus examination

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Cornea and Cataract Consultants of Arizona, Phoenix, Arizona
  - Global Research Management, Glendale, California
  - North Bay Eye Associates, Inc., Petaluma, California
  - ICON Eye Care, Grand Junction, Colorado
  - Comprehensive Eye Care, Ltd., Washington, Missouri
  - Cincinnati Eye Institute - Blue Ash, Blue Ash, Ohio